CLINICAL TRIAL: NCT06941142
Title: An Ib/III Study to Evaluate the Safety and Efficacy of Sirolimus（Albumin-bound）in Combination With Palbociclib and Fulvestrant in Patients With Advanced HR- Positive, HER2- Negative Breast Cancer
Brief Title: A Study of Sirolimus (Albumin-Bound) in Combination With Palbociclib and Fulvestrant for the Treatment of Advanced Breast Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HB1901-009
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — Sirolimus; palbociclib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation and expansion (Experimental)
  Interventions: Drug: Sirolimus (albumin - bound); Drug: Palbociclib tablet; Drug: Fulvestrant injection

INTERVENTIONS:
Drug: Sirolimus (albumin - bound) — Dose escalation, intravenous infusion
Drug: Palbociclib tablet — The dosage is 125 mg, orally once a day. Taken continuously for three weeks followed by a one - week break, with a treatment cycle of four weeks
Drug: Fulvestrant injection — The dosage is 500 mg, intramuscular injection. It is given on the 1st and 15th days of the first cycle, with a treatment cycle of four weeks. After that, it is administered once every four weeks.

SUMMARY:
This study adopts multicenter/randomized trial design. It plans to enroll patients with HR- positive, HER2- negative advanced breast cancer who are resistant to (neo)adjuvant endocrine therapy. Dose-escalation and dose-expansion studies will be carried out to evaluate the safety, tolerability, and preliminary efficacy of sirolimus (albumin-bound) in combination with palbociclib and fulvestrant in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects should be over 18 years old, regardless of gender.
* 2. Histologically or cytologically confirmed HR - positive, HER2 - negative advanced breast cancer.
* 3. For patients in the dose escalation stage, there are no limitation on previous treatments. The investigator must assess whether the patients are currently suitable for enrollment and eligible to receive the study drug treatment. For patients in the dose expansion stage need to meet the following criteria: The patient has received (neo)adjuvant endocrine therapy and has evidence of radiographic recurrence or progression during the treatment or within 12 months after the end of the treatment. The patient is allowed to receive no more than one line of systemic chemotherapy at the recurrence and metastasis setting. The patient has not received CDK4/6 inhibitor treatment at the recurrence and metastasis setting.
* 4. At least one measurable lesion meeting RECIST V1.1 criteria (patients with bone-only metastases may be enrolled in the dose escalation stage).
* 5. The Eastern Cooperative Oncology Group (ECOG) performance status score is 0 - 1.
* 6. The predicted survival time is more than 6 months.
* 7. The major organ functions must meet the protocol criteria within 7 days prior to treatment.
* 8. Voluntarily participate in this clinical study, understand the research procedures, and be able to sign the written informed consent form.

Exclusion Criteria:

* 1. Previously diagnosed with HER2 - positive breast cancer through pathological examination.
* 2. Patients deemed by the investigator as unsuitable for endocrine therapy (e.g., those with visceral crisis posing immediate life-threatening risks in the short term, including: uncontrolled massive effusions [pleural, pericardial, or peritoneal], pulmonary lymphangitic carcinomatosis, or hepatic involvement >50%).
* 3. Patients who have previously received treatment with fulvestrant or inhibitors such as PI3K/AKT/mTOR.
* 4. Patients with uncontrolled third-space fluid accumulation (e.g., pericardial effusion, pleural effusion, or ascites) requiring repeated drainage or other therapeutic interventions, and deemed ineligible for enrollment by investigators.
* 5. Patients with a history of severe lung diseases, such as interstitial lung disease and/or pneumonia, or pulmonary hypertension, or radiation pneumonia requiring glucocorticoid treatment.
* 6. Patients with chronic gastrointestinal dysfunction mainly manifested as diarrhea, such as Crohn's disease, ulcerative colitis, malabsorption, or diarrhea of grade ≥ 1; intestinal obstruction, or other gastrointestinal diseases deemed clinically significant by investigators.
* 7. Patients with known coagulation disorders such as bleeding tendency; or those who need to use anticoagulants, which may affect the intramuscular injection of fulvestrant or the use of LHRH agonists.
* 8. Patients with known hypersensitivity or intolerance to any component of the investigational drug(s), their excipients, or LHRH agonists (if applicable).
* 9. Patients with a history of autoimmune diseases (except tuberous sclerosis), immunodeficiency diseases (including positive HIV test), or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
The occurrence and frequency of adverse events (AE) | up to 2 years
dose-limiting toxicities (DLT) | up to 1 year
The recommended phase 3 dose | up to 2 years
The occurrence and frequency of serious adverse events (SAE) | up to 2 years
Overall reponse rate（ORR） | up to 2 years